CLINICAL TRIAL: NCT05936190
Title: Comparison of the Effect of Lidocaine Infusion Applied at Different Doses During Lumbar Spinal Surgery on Hemodynamics and Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Collaborators: Dilek Yörükoğlu (Unknown); Ozan Uyan (Unknown)
Responsible Party: Principal Investigator, Süheyla Karadağ Erkoç, Anesthesiology and Reanimation, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: AnkaraULumbarSurgeryLidocaine
Record Dates: First submitted 2023-03-23; First posted 2023-07-07 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Post Operative Pain; Hemodynamic Instability; Opioid Use
Keywords: lidocaine; infusion; postoperative pain; lumbar surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group L1 (Active Comparator): Group who gets 1 mg/kg/min IV lidocaine infusion during surgery
  Interventions: Drug: Lidocaine
- Group L2 (Experimental): Group who gets 2 mg/kg/min IV lidocaine infusion during surgery
  Interventions: Drug: Lidocaine IV

INTERVENTIONS:
Drug: Lidocaine IV — Intravenous infusion rate of lidocaine is 2 mg/kg/min
  Arms: Group L2
Drug: Lidocaine — Intravenous infusion rate of lidocaine is 1 mg/kg/min
  Arms: Group L1

SUMMARY:
The aim of this study is to investigate the effects of intravenous infusion of lidocaine at different doses (1 mg/kg/h vs. 2 mg/kg/h) in the intraoperative period in patients undergoing lumbar stabilization, whether postoperative pain, postoperative opioid use, opioid-related side effects are reduced, and its effects on intraoperative hemodynamics

DETAILED DESCRIPTION:
Lumbar stabilization surgery is among the surgical interventions with a high incidence of postoperative pain. Controlling postoperative pain and ensuring early recovery are important in terms of early neurological evaluation. It has been shown that lidocaine infusion administered during the intraoperative period causes peripheral vasodilation, synaptic transmission inhibition, and an increase in the depth of anesthesia. Because of these effects, the effects of lidocaine infusion on hemodynamic responses and recovery have been investigated. The safe dose range of lidocaine is 1-4 mg/kg, and the toxic dose is 5 mg/kg and above. Many studies have shown that lidocaine infusion suppresses the sympathetic reflex response and has a depressive effect on the cardiovascular system. In a study evaluating patients who underwent open radical prostatectomy surgery, it was found that blood pressure values were lower in patients who received intraoperative lidocaine infusion compared to the control group. In a study evaluating 60 female patients who underwent breast surgery, it was shown that the mean blood pressure value was significantly lower in patients who received lidocaine infusion. Lidocaine infusion has been applied at different doses (2-3 mg/kg/hour) and at different times in different surgical procedures, and it has been shown to be more effective in reducing postoperative pain, especially in some surgical procedures. Studies showing that lidocaine infusion provides early recovery in the perioperative period; They explain this effect of lidocaine by reducing the need for opioids and reducing the complications that affect the quality of recovery, such as opioid-related nausea and vomiting. It has been shown that 2 mg/kg/hour lidocaine infusion in patients undergoing vertebral surgery provides early and high-quality recovery by reducing the opioid requirement and reducing pain scores. In a study conducted in patients undergoing spinal fusion surgery, lidocaine was administered as a bolus of 2 mg/kg in the induction of anesthesia and infusion of 3 mg/kg/hour in the intraoperative period until the end of the surgery. Compared to the control group, the first additional analgesic need emerged later and the total amount of morphine consumption was found to be lower. Although there are studies in the literature using different doses of lidocaine in different surgeries, there are limited data on the effect of different doses of lidocaine on intraoperative postoperative pain and hemodynamics in patients who underwent vertebral surgery. In our study, we aimed to investigate the effect of different doses of lidocaine infusion (1 mg/kg/hour and 2 mg/kg/hour) on postoperative pain changes and hemodynamics. The main aim of the study is to evaluate whether 2 mg/kg/h lidocaine infusion doses reduce postoperative pain severity more than 1 mg/kg/h infusion doses in patients undergoing lumbar stabilization surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1,2

Exclusion Criteria:

* ASA 3,4,5
* Pediatric Patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Assessing Postoperative pain with the pain scoring system (Visual Pain Scale). | 24 hours
  The primary endpoint was the evaluation and comparison of two different infusion doses (2 mg/kg/hr and 1 mg/kg/hr) of postoperative pain with the pain scoring system (Visual Pain Scale).

SECONDARY OUTCOMES:
Monitoring Intraoperative blood pressure | 2 hours
  The secondary endpoint was to determine and compare the effect of two different infusion doses on intraoperative blood pressure
Monitoring intraoperative heart rate | 2 hours
  The secondary endpoint was to determine and compare the effect of two different infusion doses on intraoperative heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Abou-Madi MN, Keszler H, Yacoub JM. Cardiovascular reactions to laryngoscopy and tracheal intubation following small and large intravenous doses of lidocaine. Can Anaesth Soc J. 1977 Jan;24(1):12-9. doi: 10.1007/BF03006808. PMID 832175
- [Result] Weibel S, Jelting Y, Pace NL, Helf A, Eberhart LH, Hahnenkamp K, Hollmann MW, Poepping DM, Schnabel A, Kranke P. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery in adults. Cochrane Database Syst Rev. 2018 Jun 4;6(6):CD009642. doi: 10.1002/14651858.CD009642.pub3. PMID 29864216
- [Result] Saadawy IM, Kaki AM, Abd El Latif AA, Abd-Elmaksoud AM, Tolba OM. Lidocaine vs. magnesium: effect on analgesia after a laparoscopic cholecystectomy. Acta Anaesthesiol Scand. 2010 May;54(5):549-56. doi: 10.1111/j.1399-6576.2009.02165.x. Epub 2009 Nov 16. PMID 19919581
- [Result] Koshyari HS, Asthana V, Agrawal S. Evaluation of lignocaine infusion on recovery profile, quality of recovery, and postoperative analgesia in patients undergoing total abdominal hysterectomy. J Anaesthesiol Clin Pharmacol. 2019 Oct-Dec;35(4):528-532. doi: 10.4103/joacp.JOACP_209_18. PMID 31920239
- [Result] Ibrahim A, Aly M, Farrag W. Effect of intravenous lidocaine infusion on long-term postoperative pain after spinal fusion surgery. Medicine (Baltimore). 2018 Mar;97(13):e0229. doi: 10.1097/MD.0000000000010229. PMID 29595671
- [Result] Weinberg L, Jang J, Rachbuch C, Tan C, Hu R, McNicol L. The effects of intravenous lignocaine on depth of anaesthesia and intraoperative haemodynamics during open radical prostatectomy. BMC Res Notes. 2017 Jul 6;10(1):248. doi: 10.1186/s13104-017-2570-4. PMID 28683817
- [Result] Choi SJ, Kim MH, Jeong HY, Lee JJ. Effect of intraoperative lidocaine on anesthetic consumption, and bowel function, pain intensity, analgesic consumption and hospital stay after breast surgery. Korean J Anesthesiol. 2012 May;62(5):429-34. doi: 10.4097/kjae.2012.62.5.429. Epub 2012 May 24. PMID 22679539